CLINICAL TRIAL: NCT01235494
Title: Development of New MRI Pulse Sequences for Probing Lung Function in Volunteers With Hyperpolarised 3He Gas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STH15080
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- polarised 3 helium (Experimental): inhaled gas
  Interventions: Other: polarised 3 helium

INTERVENTIONS:
Other: polarised 3 helium — 1 inhalation (= 1 litre)

SUMMARY:
To develop techniques with MRI of Helium-3 gas to give functional images of the lungs. The goal is to test a single breath-hold functional 3-He MRI pulse sequence with sensitivity to multiple functional aspects of the luncg physiology. A group of 20 healthy volunteers willbe recruited from the local research group and the results compared with existing methods that require seperate breath-holds of 3He gas

ELIGIBILITY:
Inclusion Criteria:

* age 18 -70

Exclusion Criteria:

* contraindication to MRI
* Resting oxygen saturation <95%
* Volunteers requiring bronchodilators less than 4 hourly
* additional respiratory diagnoses
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Unit of Radiology, Univeristy of Sheffield, Sheffield, South Yorkshire, United Kingdom